CLINICAL TRIAL: NCT07157800
Title: Effectiveness of Exercises Given Along With Ergonomics Training in Construction Workers: A Randomized Controlled Trial
Brief Title: Effectiveness of Exercises Given Along With Ergonomics Training in Construction Workers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Doç.Dr.Ömer Şevgin, Assoc.Prof.Dr., Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Uskudar100
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Work-related Illness
MeSH Terms: interventions — Ergonomics; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): control group
  Interventions: Other: ergonomics training
- exercise group (Experimental): exercise group
  Interventions: Other: ergonomics training; Other: exercise + ergonomics training

INTERVENTIONS:
Other: ergonomics training — Each of the control group participants will receive separate ergonomics training. The content of this training will include the topics of "what is ergonomics, the purpose of ergonomics, musculoskeletal diseases in employees, work-related musculoskeletal risk factors.
Other: exercise + ergonomics training — Each of the control group participants will receive separate ergonomics training. The content of this training will include the topics of "what is ergonomics, the purpose of ergonomics, musculoskeletal diseases in employees, work-related musculoskeletal risk factors.
  Other: exercise program stretching exercises strengthening exercises waist exercises core exercises relaxation exercises
  Arms: exercise group

SUMMARY:
This research aims to examine the effectiveness of exercises given along with ergonomics training in construction workers.

DETAILED DESCRIPTION:
The study is a randomized controlled study. This study will be conducted on construction workers in the Edremit district of Balıkesir. The study will be conducted by a physiotherapist. Participants will be divided into two groups. The construction workers included in the study will be divided into an experimental group and a control group using a simple randomization method. Randomization will be conducted using a sealed envelope method. All participants will sign an informed consent form before the study begins. The assigned exercises will be monitored using an exercise tracking chart. The control group will receive only ergonomics training. The experimental group will receive both ergonomics and exercise training. Participants will receive treatment three times per week, each session lasting 45-60 minutes, for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male individuals aged 25-55
* Individuals with a visual analog scale score of ≥ 3 and a functional loss that does not completely limit their daily life
* Complaints of back, knee, neck, wrist, or shoulder pain for the last 3 months
* No surgical intervention within the last year
* Working 45 hours or more per week
* Individuals who volunteered to participate in the study and signed a written informed consent form, understanding the purpose and process of the study

Exclusion Criteria

* Presence of a respiratory system disease
* Presence of an orthopedic or neurological disease
* Presence of a psychological disorder that may affect pain perception (e.g., depression, anxiety)

Ages: 25 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-09-09 (Actual); Primary Completion 2025-12-08 (Actual); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
The Pittsburgh Sleep Quality Index | 14 weeks
  Pittsburgh Sleep Quality Index; It evaluates sleep duration, sleep disturbance, sleep efficiency, subjective sleep quality, sleep medication use, daytime dysfunction, and sleep delay and consists of a total of 24 questions. 19 of them are self-report scales and 5 of them consist of questions to be answered by a friend or spouse. There are 7 components with 18 questions scored in the scale, and each component is evaluated between 0 and 3 points. The total score ranges from 0 to 21, and 5 or more is an indicator of "poor sleep quality
Maslach Burnout Scale | 14 weeks
  The scale consists of 22 questions in total. A 5-point Likert scale is used to answer the questions. There are options such as 0- Never, 1- Rarely, 2- Sometimes, 3- Often, 4- Always. Volunteers are asked to tick the appropriate option for each question. The scale has 3 sub-categories. There are 9 items for the emotional exhaustion section, 5 items for the depersonalization section, and 8 items for the personal achievement section. People with high burnout levels are expected to have high scores on the emotional exhaustion section and depersonalization section, and low personal achievement scores. The scores that can be obtained from the subscales range from 0-36 for emotional exhaustion, 0-20 for depersonalization, and 0-32 for personal achievement.
Nordic Musculoskeletal Questionnaire | 14 weeks
  It is a scale used to determine the extent of pain in the musculoskeletal system. The purpose of this questionnaire is to identify and compare pain and complaints in parts of the body. There is an image showing the 9 parts of the body included in the questionnaire. These body parts; neck, shoulders, back, elbows, hands, waist, hips, knees and feet. The respondents are asked whether they have experienced problems such as pain and discomfort in their body parts in the last 12 months, in the last 4 weeks, and on the day of the assessment, and they are asked to mark this as yes or no.
Fatigue severity scale | 14 weeks
  The lowest score that can be obtained from the scale is 9, and the highest score is 63. The fatigue severity scale is the average value of nine sections. A high score indicates increased fatigue severity. The scale, including the day it was filled, questions the state of fatigue in the last 1 month.

CONTACTS AND LOCATIONS:
Overall Officials: Betül YILDIZ, Study Chair — Uskudar University
Locations (1):
- Building, Balıkesir, Edremit, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhao J, Obonyo E, G Bilen S. Wearable Inertial Measurement Unit Sensing System for Musculoskeletal Disorders Prevention in Construction. Sensors (Basel). 2021 Feb 13;21(4):1324. doi: 10.3390/s21041324. PMID 33668433
- [Background] Sarotto AJ, Besse M, Ambrosini L, Baldassarre R, Rosado J, Baigorria J. [Lumbosacral arthrodesis in construction workers. Return to work]. Medicina (B Aires). 2021;81(5):742-748. Spanish. PMID 34633946
- [Background] Yang F, Di N, Guo WW, Ding WB, Jia N, Zhang H, Li D, Wang D, Wang R, Zhang D, Liu Y, Shen B, Wang ZX, Yin Y. The prevalence and risk factors of work related musculoskeletal disorders among electronics manufacturing workers: a cross-sectional analytical study in China. BMC Public Health. 2023 Jan 3;23(1):10. doi: 10.1186/s12889-022-14952-6. PMID 36597111
- [Background] Lee S, Kim YJ, Kim Y, Kang D, Kim SC, Kim SY. Incidence rates of injury, musculoskeletal, skin, pulmonary and chronic diseases among construction workers by classification of occupations in South Korea: a 1,027 subject-based cohort of the Korean Construction Worker's Cohort (KCWC). Ann Occup Environ Med. 2023 Jul 24;35:e26. doi: 10.35371/aoem.2023.35.e26. eCollection 2023. PMID 37614337